CLINICAL TRIAL: NCT04163081
Title: The INITIATE Study: Initiating Nicotine Dependence Treatment for Smokers Admitted to Emergency Departments
Acronym: INITIATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20190485-01H
Record Dates: First submitted 2019-10-07; First posted 2019-11-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-10

CONDITIONS: Nicotine Dependence, Cigarettes; Nicotine Withdrawal
Keywords: Nicotine Replacement Therapy; Emergency Department; Nicotine Dependence; Tobacco Abstinence; Tobacco Treatment; Cigarette
MeSH Terms: conditions — Tobacco Use Disorder; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quit Card Intervention (QCI) (Experimental): Study intervention group.
  Interventions: Behavioral: Quit Card Intervention (QCI)
- Usual Care (UC) (No Intervention): Study control group.

INTERVENTIONS:
Behavioral: Quit Card Intervention (QCI) — The intervention is comprised of a behavioural incentive in the form of a gift card as well as tailored smoking cessation counseling. Eligible consenting smokers randomized to the QCI group will receive: a "Quit Card" (a gift card worth $300 that can be used to buy nicotine replacement therapies at any pharmacy); self-help information; and, enrollment in six months of telephone follow-up support tailored by treatment goal with a Nicotine Addiction Treatment Specialist.
  Arms: Quit Card Intervention (QCI)

SUMMARY:
The INITIATE Study is a randomized controlled trial that is testing an intervention designed to increase long-term abstinence among tobacco smokers seen in emergency departments (ED) and other high-volume hospital and community ambulatory care settings. The intervention includes a behavioural incentive and tailored follow-up support on long-term smoking abstinence, health, healthcare utilization, and cost. Tobacco-related illnesses cost the healthcare system millions each year. Quitting smoking improves smoking-related outcomes, like the onset or management of heart disease, stroke, lung diseases, and several cancers. There are approximately 16 million visits to Canadian EDs each year; an estimated 3-4 million of these involve smokers. Effective quit smoking interventions exist, but are underutilized. Few hospital EDs, community healthcare centers, and other inpatient and outpatient clinics in Canada offer tobacco-use interventions. In order for clinicians to offer quit smoking support, interventions need to be simple given the realities of these high-volume environments. Considering that stopping smoking improves health outcomes, that tobacco-use is an important cause of preventable ED use, and the volume of smokers, Canadian EDs and other high-volume hospital and community ambulatory care settings are a missed opportunity in the initiation of quit smoking support. Our intervention has been designed to optimize uptake and smoking abstinence by including the most effective evidence-based behavioural and drug-related approaches, removing specific barriers and challenges that smokers face when trying to quit (e.g., affordability, low confidence and motivation), while packaging the intervention in a quick-to-initiate manner, making it ideal for fast-paced, complex environments.

ELIGIBILITY:
Inclusion Criteria:

* Current daily smoker (smokes ≥ 5 cigarettes per day);
* ≥ 18 years of age (the age of majority in Ontario);
* For ED sites only, assigned a CTAS level of 2-5 (emergent to non-urgent);
* Able to read and understand English or French;
* Resides in Ontario and eligible for Ontario Health Insurance Plan (to permit linkage with administrative data housed at the Institute for Clinical Evaluative Sciences [ICES]);
* Available and willing to participate in follow-up assessments over the next 12 months;
* Has access to a telephone or computer;
* Able to provide informed consent

Exclusion Criteria:

* Currently participating in this or another smoking cessation study;
* For ED sites only, assigned a CTAS level of 1 (resuscitation - the most seriously ill patients with highest likelihood of hospital admission) or in psychiatric emergency unit;
* Pregnant, planning to become pregnant over the next year, or breastfeeding;
* Has morbid illness which will prevent completion of 26-week follow-up (e.g., receiving palliative care);
* In the opinion of the attending physician, manifests acute physical and/or psychiatric illness or has cognitive impairment that would preclude participation in/benefit from the intervention.
* Scheduled for a known elected surgery, procedure, or future hospitalization during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1208 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Smoking Abstinence | 26 weeks (6 months) after study enrollment
  Smoking abstinence at 26 weeks, biochemically verified using an expired air carbon monoxide (CO) test

SECONDARY OUTCOMES:
Prolonged Abstinence | 4, 26, and 52 weeks after study enrollment
  Prolonged (since last time point) smoking abstinence, at 4, 26, and 52 weeks
Point Prevalence Abstinence | 4, and 52 weeks after study enrollment
  Point prevalence smoking abstinence, at 4, and 52 weeks
Smoking Reduction | 4, 26, and 52 weeks after study enrollment
  Smoking reduction (i.e., change in number of daily cigarettes), at 4, 26, and 52 weeks
Number of Quit Attempts | 4, 26, and 52 weeks after study enrollment
  Number of quit attempts since study entry, at 4, 26, and 52 weeks
Cessation Medication and/or E-cigarette Use | 4, 26, and 52 weeks after study enrollment
  Use of smoking cessation medication and/or e-cigarette, at 4, 26, and 52 weeks
Use of Behavioural Supports | 4, 26, and 52 weeks after study enrollment
  Use of behavioural supports (e.g., counseling, quit lines), at 4, 26, and 52 weeks
Health-Related Quality of Life | 52 weeks after study enrollment
  Health-related quality of life (HR-QoL), at 52 weeks. This will be measured using the Hospital Anxiety and Depression Scale (HADS), designed to identify and measure the levels of anxiety and depression among individuals in non-psychiatric hospital settings, and the Health Questionnaire Assessment (EQ-5D-5L), using five graded severity levels to summarize perceived health across five foundational dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Health Services Outcomes - ED visits | 4, 26, and 52 weeks after study enrollment
  Number of all-cause and smoking-related (e.g., vascular, respiratory, cancer-related) visits to ED at 4, 26, and 52 weeks
Health Services Outcomes - Hospital Admissions | 4, 26, and 52 weeks after study enrollment
  Number of all-cause and smoking-related (e.g., vascular, respiratory, cancer-related) admissions to hospital at 4, 26, and 52 weeks
Health Services Outcomes - Deaths | 4, 26, and 52 weeks after study enrollment
  Number of all-cause and smoking-related (e.g., vascular, respiratory, cancer-related) deaths at 4, 26, and 52 weeks
Cost-Effectiveness Ratios | 52 weeks after study enrollment
  Cost-effectiveness ratios related to health services at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kerri-Anne Mullen, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (4):
- Canada (4):
  - Civic Hospital, Ottawa, Ontario
  - General Hospital, Ottawa, Ontario
  - Riverside Hospital, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mullen KA, Garg A, Gagnon F, Wells G, Kapur A, Hawken S, Pipe AL, Walker K, Thiruganasambandamoorthy V, Klepaczek M, Reid RD. The INITIATE trial protocol: a randomized controlled trial testing the effectiveness of a "quit card" intervention on long-term abstinence among tobacco smokers presenting to the emergency department. Trials. 2021 Oct 23;22(1):733. doi: 10.1186/s13063-021-05693-9. PMID 34688291